CLINICAL TRIAL: NCT05136651
Title: Clinical Trial of OurRelationship, a Scalable Digital Intervention for Veteran Couples
Brief Title: OurRelationship for Veteran Couples
Acronym: VA-OR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3777-W
Record Dates: First submitted 2021-11-15; First posted 2021-11-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Relationship Distress
Keywords: couples; OurRelationship; relationship; couples therapy

STUDY DESIGN:
Intervention Model Description: Waitlist-control design. Participants will be randomly assigned to receive either immediate treatment or treatment after a 2-month waiting period. The intervention received is the same in both conditions; only the timing differs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Treatment (Experimental): Couples assigned to the Immediate Treatment condition will begin the OurRelationship program immediately following random assignment.
  Interventions: Behavioral: OurRelationship
- Waitlist Control (Other): Couples assigned to the Waitlist Control condition will begin the OurRelationship program following a 2-month delay after random assignment.
  Interventions: Behavioral: OurRelationship

INTERVENTIONS:
Behavioral: OurRelationship — The OurRelationship Program is an online adaptation of Integrative Behavioral Couple Therapy (IBCT). It consists of 3 modules that couples complete over the course of 6-8 weeks. Couples also receive a 30-minute coaching appointment following completion of each module.

SUMMARY:
Access to a flexible spectrum of family-based VA mental health care for Veterans is mandated by law. Research shows that relationship distress harms Veterans' mental health, physical health, and mortality, while healthy relationships provide resilience and facilitate recovery from illness. However, there are many barriers to accessing couple and family care within VA, including system-level barriers such as insufficient access to specialty providers and couple-level barriers such as difficulty coordinating schedules and finding childcare. OurRelationship is an evidence-based, coached online intervention for couples that provides flexible, accessible, and scalable treatment to improve relationship functioning. This proposed CDA-2 project will test whether OurRelationship is effective for improving Veterans' intimate relationships and supporting their rehabilitation. This study supports the mission of the 2018-2024 Strategic Plan of the Department of Veterans Affairs by improving Veterans' relationship functioning to enhance their overall quality of life.

DETAILED DESCRIPTION:
Over 75% of Veterans referred for behavioral health assessments endorse significant relationship concerns, including 60% reporting mild to severe intimate partner violence. Relationship problems increase risk of cardiovascular illness, exacerbate psychiatric symptoms, impair social and work functioning, and are the most common precipitants of suicidal ideation and attempts for Veterans. Healthy intimate relationships are a crucial part of wellness, resilience, and recovery, and biopsychosocial theories of rehabilitation psychology stress the importance of relationships. Military Veterans have experienced numerous stressors that increase risk of relationship distress, including deployment and reintegration cycles, frequent relocation, and physical and mental health sequelae of trauma. Accordingly, VHA directive 1163.04 in 2019 mandated that all Veterans have access to a flexible continuum of family mental health services as part of rehabilitation efforts.

However, access to couples' interventions is limited, and traditional couple psychotherapy is not sufficiently scalable. Although most VA medical centers have trained couple therapists, they are limited in number and location, and they are underutilized due to numerous logistical barriers couples face including coordinating schedules, dual time off work, childcare, and stigma. Unsurprisingly, over 60% of divorced couples never accessed couples' treatment, and Veterans spend four to seven years in relationship distress before getting help. Digital health is a critical part of solving problems of access to care. Because digital health interventions for couples can provide flexible access to evidence-based relationship interventions, they are an essential part of providing the continuum of family mental health care mandated by VHA.

OurRelationship is an online adaptation of Integrative Behavioral Couple Therapy (IBCT), the evidence-based protocol for couple therapy currently in use in the VA healthcare system. It combines eight hours of a self-paced online couples' program with three 20-minute telehealth coaching sessions. OurRelationship is a scalable, transdiagnostic, evidence-based couples' intervention that can help provide access to flexible family mental health services. Several RCTs demonstrate OurRelationship improves both relationship functioning and individual mental health. A small secondary analysis from an RCT supports the use of OurRelationship with Veterans in the community, and the pilot data from 13 couples recruited over two months in the VA San Diego Healthcare System (VASDHS) indicate that Veterans find OurRelationship appealing and helpful. However, OurRelationship has not yet been empirically evaluated with a Veteran population in a VA care setting.

The scientific goals of this CDA-2 project are to evaluate the feasibility, acceptability, and efficacy of OurRelationship for improving relationship and individual functioning among Veteran couples. The proposed 5-year study is a 2-month waitlist-controlled randomized clinical trial. The investigators aim to serve 90 couples (Veterans and their partners, N = 180) who report relationship distress, recruited from mental health clinics within VASDHS. The sample and recruitment plan is feasible based on the investigators' pilot testing and on prior RCTs. Data on outcomes including relationship functioning and behavior (e.g., communication, conflict), individual functioning (e.g., quality of life, family role), and psychiatric symptoms (depression, anxiety) will be collected at baseline, mid-program, post-program, and a 6-month follow-up. The investigators will collect participant feedback via semi-structured interviews and ratings of program satisfaction and therapeutic alliance.

The Specific Aims are:

Aim 1: To examine feasibility and acceptability of implementing OurRelationship in a VA setting with Veterans and their partners, evidenced by quantitative (recruitment, retention, and satisfaction ratings) and qualitative data (semi-structured interviews soliciting participant feedback).

Aim 2: To evaluate efficacy of the OurRelationship program for Veterans and their partners, as evidenced by statistically and clinically significant improvements in relationship and individual functioning that are maintained for 6 months post-intervention.

Aim 3: To explore mediation of improvements in individual functional outcomes by improvements in relationship functioning.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be couples consisting of a Veteran referred from a mental health care clinic at VA San Diego Healthcare System and their spouse or romantic partner who is willing to participate
* Couples must:

  * both speak, read, and write English
  * be married, living together, or in a relationship for at least 12 months
  * endorse clinically significant relationship distress by one or both partner's reports (i.e., < 104.5 on the Couples Satisfaction Index-32)
  * have internet access sufficient to complete the online program and attend telehealth visits
  * be willing to have telehealth coach sessions audio-recorded

Exclusion Criteria:

* Couples will be excluded if either partner reports

  * an active substance use disorder within the past three months (i.e., 2+ on the TAPS screening tool for a single substance followed by positive diagnosis in clinical interview)
  * a diagnosis of a psychotic or bipolar disorder with current uncontrolled symptoms (by self-report)
  * a diagnosis of severe cognitive impairment or intellectual disability (by self-report)
  * severe physical or sexual relationship aggression during the past 12 months (i.e., 10+ on the Hurt-Insult-Threaten-Scream [HITS] screening tool followed by clinical interview)
  * current suicidal ideation or behavior determined to be high-risk according to current VA clinical assessment protocols (i.e., "yes" on any high-risk items on the Columbia Suicide Severity Rating Scale)
  * suicide-related hospitalizations within the past 12 months (by self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Couples Satisfaction Index (CSI-32) | Baseline
  The Couples Satisfaction Index (CSI-32) is a 32-item measure designed to assess relationship satisfaction of intact (married, cohabiting or dating) couples. The measure includes items aimed at assessing the presence of problems between individuals and the intensity of such problems. Total scores can range from 0 to 161. Higher scores indicate higher levels of relationship satisfaction. CSI-32 scores falling below 104.5 suggest clinical relationship distress.
Couples Satisfaction Index (CSI-32) | Mid-treatment (approx. 1 month post-randomization)
  The Couples Satisfaction Index (CSI-32) is a 32-item measure designed to assess relationship satisfaction of intact (married, cohabiting or dating) couples. The measure includes items aimed at assessing the presence of problems between individuals and the intensity of such problems. Total scores can range from 0 to 161. Higher scores indicate higher levels of relationship satisfaction. CSI-32 scores falling below 104.5 suggest clinical relationship distress.
Couples Satisfaction Index (CSI-32) | Post-treatment (approx. 2 months post-randomization)
  The Couples Satisfaction Index (CSI-32) is a 32-item measure designed to assess relationship satisfaction of intact (married, cohabiting or dating) couples. The measure includes items aimed at assessing the presence of problems between individuals and the intensity of such problems. Total scores can range from 0 to 161. Higher scores indicate higher levels of relationship satisfaction. CSI-32 scores falling below 104.5 suggest clinical relationship distress.
Couples Satisfaction Index (CSI-32) | 6-month follow-up (approx. 6 months following completion of post-treatment assessment)
  The Couples Satisfaction Index (CSI-32) is a 32-item measure designed to assess relationship satisfaction of intact (married, cohabiting or dating) couples. The measure includes items aimed at assessing the presence of problems between individuals and the intensity of such problems. Total scores can range from 0 to 161. Higher scores indicate higher levels of relationship satisfaction. CSI-32 scores falling below 104.5 suggest clinical relationship distress.

SECONDARY OUTCOMES:
Depression, Anxiety, and Stress Scale (DASS-21) | 6-month follow-up (approx. 6 months following completion of post-treatment assessment)
  Psychological distress will be measured with the Depression, Anxiety, and Stress Scale (DASS-21), a 21-item self-report questionnaire measuring three dimensions of negative emotional states. Each of the three dimensions is measured with 7 items on a 0 to 3 point scale, and total scores are calculated by summing the items and then doubling the sum score for equivalence to the longer DASS-42. Total scores for the three dimensions range from 0 to 42.
Communication Skills Test (CST-10) | Baseline
  Positive communication will be measured using the Communication Skills Test (CST), a 10-item assessment of self-reported use of adaptive communication skills (e.g., paraphrasing, time-out). Responses use a 7-point Likert-type scale and are averaged to range from 0 to 7, with higher scores representing better communication skills.
Communication Skills Test (CST-10) | Mid-treatment (approx. 1 month post-randomization)
  Positive communication will be measured using the Communication Skills Test (CST), a 10-item assessment of self-reported use of adaptive communication skills (e.g., paraphrasing, time-out). Responses use a 7-point Likert-type scale and are averaged to range from 0 to 7, with higher scores representing better communication skills.
Communication Skills Test (CST-10) | Post-treatment (approx. 2 months post-randomization)
  Positive communication will be measured using the Communication Skills Test (CST), a 10-item assessment of self-reported use of adaptive communication skills (e.g., paraphrasing, time-out). Responses use a 7-point Likert-type scale and are averaged to range from 0 to 7, with higher scores representing better communication skills.
Communication Skills Test (CST-10) | 6-month follow-up (approx. 6 months following completion of post-treatment assessment)
  Positive communication will be measured using the Communication Skills Test (CST), a 10-item assessment of self-reported use of adaptive communication skills (e.g., paraphrasing, time-out). Responses use a 7-point Likert-type scale and are averaged to range from 0 to 7, with higher scores representing better communication skills.
Communication Danger Signs Scale (CDS) | Baseline
  Negative communication will be measured using the Communication Danger Signs scale (CDS), an 8-item scale assessing specific negative communication behaviors that are associated with relationship dissolution. Responses use a 7-point Likert-type scale and are averaged to range from 0 to 7, with higher scores representing more negative communication.
Communication Danger Signs Scale (CDS) | Mid-treatment (approx. 1 month post-randomization)
  Negative communication will be measured using the Communication Danger Signs scale (CDS), an 8-item scale assessing specific negative communication behaviors that are associated with relationship dissolution. Responses use a 7-point Likert-type scale and are averaged to range from 0 to 7, with higher scores representing more negative communication.
Communication Danger Signs Scale (CDS) | Post-treatment (approx. 2 months post-randomization)
  Negative communication will be measured using the Communication Danger Signs scale (CDS), an 8-item scale assessing specific negative communication behaviors that are associated with relationship dissolution. Responses use a 7-point Likert-type scale and are averaged to range from 0 to 7, with higher scores representing more negative communication.
Communication Danger Signs Scale (CDS) | 6-month follow-up (approx. 6 months following completion of post-treatment assessment)
  Negative communication will be measured using the Communication Danger Signs scale (CDS), an 8-item scale assessing specific negative communication behaviors that are associated with relationship dissolution. Responses use a 7-point Likert-type scale and are averaged to range from 0 to 7, with higher scores representing more negative communication.
Revised Conflict Tactics Scale, Short Form (CTS-2S) | Baseline
  Conflict/aggression will be measured using the Revised Conflict Tactics Scale (CTS-2), a 20-item measure of 5 domains of relationship conflict and aggression perpetrated by the respondent and their partner. Respondents report how often each event occurred during the past month on a scale from 0 (never) to 6 (more than 20 times) Each domain is scored separately using either sum scores ranging from 0 to 24, chronicity scores ranging from 1 to 80, or prevalence scores ranging from 0 to 1.
Revised Conflict Tactics Scale, Short Form (CTS-2S) | Mid-treatment (approx. 1 month post-randomization)
  Conflict/aggression will be measured using the Revised Conflict Tactics Scale (CTS-2), a 20-item measure of 5 domains of relationship conflict and aggression perpetrated by the respondent and their partner. Respondents report how often each event occurred during the past month on a scale from 0 (never) to 6 (more than 20 times) Each domain is scored separately using either sum scores ranging from 0 to 24, chronicity scores ranging from 1 to 80, or prevalence scores ranging from 0 to 1.
Revised Conflict Tactics Scale, Short Form (CTS-2S) | Post-treatment (approx. 2 months post-randomization)
  Conflict/aggression will be measured using the Revised Conflict Tactics Scale (CTS-2), a 20-item measure of 5 domains of relationship conflict and aggression perpetrated by the respondent and their partner. Respondents report how often each event occurred during the past month on a scale from 0 (never) to 6 (more than 20 times) Each domain is scored separately using either sum scores ranging from 0 to 24, chronicity scores ranging from 1 to 80, or prevalence scores ranging from 0 to 1.
Revised Conflict Tactics Scale, Short Form (CTS-2S) | 6-month follow-up (approx. 6 months following completion of post-treatment assessment)
  Conflict/aggression will be measured using the Revised Conflict Tactics Scale (CTS-2), a 20-item measure of 5 domains of relationship conflict and aggression perpetrated by the respondent and their partner. Respondents report how often each event occurred during the past month on a scale from 0 (never) to 6 (more than 20 times) Each domain is scored separately using either sum scores ranging from 0 to 24, chronicity scores ranging from 1 to 80, or prevalence scores ranging from 0 to 1.
Brief Inventory of Psychosocial Functioning (B-IPF) | Baseline
  Psychosocial functioning will be measured using the Brief Inventory of Psychosocial Functioning (B-IPF), a 7-item measure assessing seven domains of overall functioning. Scores are calculated as percentages and range from 0 to 100, with higher scores indicating more psychosocial dysfunction (i.e., worse psychosocial functioning).
Brief Inventory of Psychosocial Functioning (B-IPF) | Mid-treatment (approx. 1 month post-randomization)
  Psychosocial functioning will be measured using the Brief Inventory of Psychosocial Functioning (B-IPF), a 7-item measure assessing seven domains of overall functioning. Scores are calculated as percentages and range from 0 to 100, with higher scores indicating more psychosocial dysfunction (i.e., worse psychosocial functioning).
Brief Inventory of Psychosocial Functioning (B-IPF) | Post-treatment (approx. 2 months post-randomization)
  Psychosocial functioning will be measured using the Brief Inventory of Psychosocial Functioning (B-IPF), a 7-item measure assessing seven domains of overall functioning. Scores are calculated as percentages and range from 0 to 100, with higher scores indicating more psychosocial dysfunction (i.e., worse psychosocial functioning).
Brief Inventory of Psychosocial Functioning (B-IPF) | 6-month follow-up (approx. 6 months following completion of post-treatment assessment)
  Psychosocial functioning will be measured using the Brief Inventory of Psychosocial Functioning (B-IPF), a 7-item measure assessing seven domains of overall functioning. Scores are calculated as percentages and range from 0 to 100, with higher scores indicating more psychosocial dysfunction (i.e., worse psychosocial functioning).
Brunnsviken Brief Quality of life scale (BBQ) | Baseline
  The Brunnsviken Brief Quality of life scale (BBQ) measures subjective quality of life validated for use with both clinical and non-clinical samples, forming an overall life satisfaction score comprised of six life domains (Leisure time, View on life, Creativity, Learning, Friends and Friendship, and View of self) assessed with two items each (importance and satisfaction). Scores are calculated by summing the products of the satisfaction and importance scores for each domain. Sum scores can range from 0 to 96, with higher scores indicating better quality of life.
Brunnsviken Brief Quality of life scale (BBQ) | Mid-treatment (approx. 1 month post-randomization)
  The Brunnsviken Brief Quality of life scale (BBQ) measures subjective quality of life validated for use with both clinical and non-clinical samples, forming an overall life satisfaction score comprised of six life domains (Leisure time, View on life, Creativity, Learning, Friends and Friendship, and View of self) assessed with two items each (importance and satisfaction). Scores are calculated by summing the products of the satisfaction and importance scores for each domain. Sum scores can range from 0 to 96, with higher scores indicating better quality of life.
Brunnsviken Brief Quality of life scale (BBQ) | Post-treatment (approx. 2 months post-randomization)
  The Brunnsviken Brief Quality of life scale (BBQ) measures subjective quality of life validated for use with both clinical and non-clinical samples, forming an overall life satisfaction score comprised of six life domains (Leisure time, View on life, Creativity, Learning, Friends and Friendship, and View of self) assessed with two items each (importance and satisfaction). Scores are calculated by summing the products of the satisfaction and importance scores for each domain. Sum scores can range from 0 to 96, with higher scores indicating better quality of life.
Brunnsviken Brief Quality of life scale (BBQ) | 6-month follow-up (approx. 6 months following completion of post-treatment assessment)
  The Brunnsviken Brief Quality of life scale (BBQ) measures subjective quality of life validated for use with both clinical and non-clinical samples, forming an overall life satisfaction score comprised of six life domains (Leisure time, View on life, Creativity, Learning, Friends and Friendship, and View of self) assessed with two items each (importance and satisfaction). Scores are calculated by summing the products of the satisfaction and importance scores for each domain. Sum scores can range from 0 to 96, with higher scores indicating better quality of life.
Family Role Performance Scale (FRPS) | Baseline
  Family role participation will be measured with the Family Role Performance Scale (FRPS), an 8-item self-report measure of the degree to which respondents fulfill expectations in two domains of family functioning (task- or relationship-oriented). The items are rated from 1 to 5, with higher sum scores (total range 8 to 40) indicating better fulfillment of family role expectations.
Family Role Performance Scale (FRPS) | Mid-treatment (approx. 1 month post-randomization)
  Family role participation will be measured with the Family Role Performance Scale (FRPS), an 8-item self-report measure of the degree to which respondents fulfill expectations in two domains of family functioning (task- or relationship-oriented). The items are rated from 1 to 5, with higher sum scores (total range 8 to 40) indicating better fulfillment of family role expectations.
Family Role Performance Scale (FRPS) | Post-treatment (approx. 2 months post-randomization)
  Family role participation will be measured with the Family Role Performance Scale (FRPS), an 8-item self-report measure of the degree to which respondents fulfill expectations in two domains of family functioning (task- or relationship-oriented). The items are rated from 1 to 5, with higher sum scores (total range 8 to 40) indicating better fulfillment of family role expectations.
Family Role Performance Scale (FRPS) | 6-month follow-up (approx. 6 months following completion of post-treatment assessment)
  Family role participation will be measured with the Family Role Performance Scale (FRPS), an 8-item self-report measure of the degree to which respondents fulfill expectations in two domains of family functioning (task- or relationship-oriented). The items are rated from 1 to 5, with higher sum scores (total range 8 to 40) indicating better fulfillment of family role expectations.
Depression, Anxiety, and Stress Scale (DASS-21) | Baseline
  Psychological distress will be measured with the Depression, Anxiety, and Stress Scale (DASS-21), a 21-item self-report questionnaire measuring three dimensions of negative emotional states. Each of the three dimensions is measured with 7 items on a 0 to 3 point scale, and total scores are calculated by summing the items and then doubling the sum score for equivalence to the longer DASS-42. Total scores for the three dimensions range from 0 to 42.
Depression, Anxiety, and Stress Scale (DASS-21) | Mid-treatment (approx. 1 month post-randomization)
  Psychological distress will be measured with the Depression, Anxiety, and Stress Scale (DASS-21), a 21-item self-report questionnaire measuring three dimensions of negative emotional states. Each of the three dimensions is measured with 7 items on a 0 to 3 point scale, and total scores are calculated by summing the items and then doubling the sum score for equivalence to the longer DASS-42. Total scores for the three dimensions range from 0 to 42.
Depression, Anxiety, and Stress Scale (DASS-21) | Post-treatment (approx. 2 months post-randomization)
  Psychological distress will be measured with the Depression, Anxiety, and Stress Scale (DASS-21), a 21-item self-report questionnaire measuring three dimensions of negative emotional states. Each of the three dimensions is measured with 7 items on a 0 to 3 point scale, and total scores are calculated by summing the items and then doubling the sum score for equivalence to the longer DASS-42. Total scores for the three dimensions range from 0 to 42.

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Post-treatment (approx. 2 months post-randomization)
  Program satisfaction will be measured using the Client Satisfaction Questionnaire (CSQ-8), an 8-item measure of client satisfaction with treatment designed for healthcare settings. Sum scores range from 8 to 32, with higher scores indicating better satisfaction with treatment services.
Working Alliance Inventory - Short Revised (WAI-SR) | Post-treatment (approx. 2 months post-randomization)
  Working alliance will be measured using the Working Alliance Inventory - Short Revised (WAI-SR), a 12-item measure of therapeutic working alliance. Sum scores range from 12 to 84, with higher scores indicating better therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Kayla C. Knopp, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Georgia Salivar E, Knopp K, Roddy MK, Morland LA, Doss BD. Effectiveness of online OurRelationship and ePREP programs for low-income military couples. J Consult Clin Psychol. 2020 Oct;88(10):899-906. doi: 10.1037/ccp0000606. PMID 33048570
- [Background] Doss BD, Knopp K, Roddy MK, Rothman K, Hatch SG, Rhoades GK. Online programs improve relationship functioning for distressed low-income couples: Results from a nationwide randomized controlled trial. J Consult Clin Psychol. 2020 Apr;88(4):283-294. doi: 10.1037/ccp0000479. PMID 32134290
- [Background] Doss BD, Cicila LN, Georgia EJ, Roddy MK, Nowlan KM, Benson LA, Christensen A. A randomized controlled trial of the web-based OurRelationship program: Effects on relationship and individual functioning. J Consult Clin Psychol. 2016 Apr;84(4):285-96. doi: 10.1037/ccp0000063. Epub 2016 Jan 25. PMID 26999504
- See also: OurRelationship Program — https://www.ourrelationship.com/